CLINICAL TRIAL: NCT03762746
Title: TMS for Treatment Resistant Auditory Verbal Hallucination in Schizophrenia
Brief Title: Transcranial Magnetic Stimulation (TMS) for Patients With Treatment Resistant Auditory Verbal Hallucination
Acronym: TMS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Khamelia Malik, Head Psychiatry Research and Development Unit, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-03-0206
Record Dates: First submitted 2018-02-23; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Hallucinations, Verbal Auditory
MeSH Terms: conditions — Hallucinations | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Forty schizophrenic or schizoaffective patients with predominant audiotoric hallucinatory symptoms will be given rTMS 1 Hz intervention, 1000-pulse train, 20 min, 90% strength, 1000 pulse in left temporo-parietal cortex for 10 consecutive days (except holidays). Assessment of DN network connectivity in the brain using the results of brain wave decomposition analysis with EEGLAB. For measurement of auditor hall of hallucinations used Indonesian-Psychosis Symptom Rating Scale (INA-PSYRATS) instrument. Source monitoring capability using the INA-Source Monitoring instrument.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: We apply blinding status of trial participants, care providers, and outcome assessors. We are using TMS sham-coil with similarities in appearance, sound, heavy; also we have the timing of final unblinding of all trial participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active (Active Comparator): Intervention with transcranial magnetic stimulation (TMS) low frequency 1 Hz , 1000-pulse train, 20 minutes, 90% motor threshold in left temporo-parietal cortex for 10 consecutive days for 20 schizophrenia patients with auditory hallucination
  Interventions: Device: Transcranial Magnetic Stimulation
- Control (Sham Comparator): Control group is received treatment as usual
  Interventions: Drug: Control

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — A custom TMS stimulator (MagStim) is used to generate repetitive biphasic magnetic pulses. Magnetic pulses are delivered with a figure-8-coil (Magnetic Coil Transducer). During the experiment, rTMS pulse intensity is adjusted to 90% of the motor threshold. Patients will be randomly assigned to receive a 1 Hz. The target area is stimulated for 10 consecutive days. Stimulation at 1 Hz was applied once a day for 10-days
  Arms: Active
Drug: Control — The control group is receiving treatment as usual. EEG recording and psychopathological ratings are performed one day before the start and on the last day of the study
  Arms: Control

SUMMARY:
This study will evaluate the effect of repetitive transcranial magnetic stimulation (rTMS) in schizophrenia with treatment resistant auditory verbal hallucination

DETAILED DESCRIPTION:
Brief summary:

This study will evaluate the effect of repetitive transcranial magnetic stimulation (rTMS) in schizophrenia with treatment resistant auditory hallucination

Detailed description:

Auditory verbal hallucinations in schizophrenia disorders have been proposed to be associated with a source- monitoring deficit. The improvement of the monitoring deficit will have major impact on the improvement of hallucinatory symptoms and the social function. Brain network considered to play a major role in source monitoring is the default mode (DM) network. An increasing activity during the brain's resting phase and decreasing activity during stimulus-induced brain activity, increased rest activity in the primary auditory cortex which contributes to conditions, internal speech perceived as a tangible external sound, triggering the occurrence of verbal auditory hallucinations in schizophrenic disorders.

This study will determine if

1-Hz low-frequency, transcranial repetitive magnetic stimulus could be used to inhibit hyperconnectivity between these DM networks and other brain regions, allowing the source-monitoring capability to function properly. This study will measure the oscillatory strength and functional connectivity in the DM network via EEG resting-state activity in schizophrenic with auditory hallucinations before and after rTMS administration. With a seed-based analysis, using the region of interest (ROIs) in the posterior cortex area of the cortex (PPC), precuneus area (PCu), the inferior parietal area (IPC), the medial temporal (MT) area, the medial frontal area (MFC) and the singulatum cortex anterior (ACC) in bilateral hemispheres to create an EEG-based brain activity mapping, measuring cortical spectral power and functional connectivity in the ROIs.

Before starting rTMS, participants will undergo : (1) general and psychiatric assessment, (2) neuropsychological test to evaluate hallucination and source-monitoring ability, (3) an EEG recording (which takes about 1 hour). After these assessment are completed, participants will be randomly assigned (by computer program) to receive either 1 Hz frequency rTMS or placebo stimulation for 20 minutes per day over a 10-day period. During this time, the participants will not know whether they received real or placebo TMS. For 10-days, stimulation will be administered to an area of the left temporal lobe of the brain (temporo-parietal junction).

After trial is completed, participants will be told if they received real or placebo. If the participants have receive only place stimulation, they will then be offered a trial of real rTMS.

TMS is not causing pain, but it can be uncomfortable due to a tingling or knocking sensation, contraction of scalp and facial muscles. There is also a small risk of seizure associated with TMS, but because of the lower frequency of stimulation used in this study (1 stimulation per second), this risk is significant only for participants who have a prior history of seizures, epilepsy, or other neurological problem. Investigators are also concerned that TMS may cause hearing problems. Therefore, investigators will carefully monitor participants for early signs of such problem, using hearing-safety aid to every stimulation session. If investigators suspect that a participant is experiencing problems with hearing, the trial is stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Met the criteria of all types of schizophrenia or schizoaffective based on structured clinical interview instruments for the DSM-IV axis I disorders (SCID-I)
2. Patients had entered the stabilization phase with 2 to 3 months of antipsychotic treatment and no drug changes within the last 2 (two) months
3. Elementary school graduated (minimum)

Exclusion Criteria:

1. Patients with a history of stroke, heart failure, head injury, infection or brain tumor, epilepsy, alcohol and opiate abuse, amphetamines obtained from anamnesis, physical examination and patient medical records
2. Patients with neurological focal deficits such as hemiparesis and cranial nerve paresis
3. Patients with severe cognitive deficits (MMSE scores <25 in the first and second graders of Senior Secondary School and <21 in Primary School Graduates)
4. Patients with severe hearing loss were assessed with a 5-word auditory test
5. Patients with mental retardation, assessed using the Wechsler Test of Adult Reading (WTAR) test and data from medical records.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Hallucinations change | 2 weeks
  Hallucinations score by Indonesia Version-Psychotic Symptom Rating Scale or PSYRATS. This auditory hallucination scale included 11 items and rated from zero to four. Symptoms over the last week will rated. The dimensions of auditory hallucinations are: frequency, duration, location, loudness, beliefs about origin, negative content, intensity of negative content, amount of distress, intensity of distress, disruption of life and control. Investigators will measure hallucination score before and after 10 session TMS. Total score consist of averaged score of dimensions. A higher score represent a worse outcome.
Source-monitoring ability | 2 weeks
  Source-monitoring score by source monitoring task performance. Participants will ask to distinguish word between 10 silent reading and 10 covert reading and 10 new non-presented word, before TMS and after 10 session TMS. Words are current Indonesian word extract from a verbal fluency task. During the test, word will be presented during 3 seconds on a computer screen.
  To evaluate the source monitoring performance, investigators will consider source attribution, corresponding to number incorrect attribution for source. Score range is between 0-20 A higher total score represents a worse outcome.

SECONDARY OUTCOMES:
electrophysiological changes | 2 weeks
  This study will investigate all frequency bands (delta, theta, alpha, beta, gamma) coherence in each region of interest of default-mode network. To examine whether functional connectivity between DMN structures differs before and after TMS, the average EEG time series for all nodes in each seed ROI will normalize using transformation and correlations will perform with all other seeds in the DMN network in a 9×9 correlation matrix. The resulting correlation coefficients for each participant will then compare using a two-sided samples t-test to evaluate between-group differences in ROI-ROI connectivity for each seed. A score will represent a functional connectivity between ROIs

CONTACTS AND LOCATIONS:
Overall Officials: Khamelia Malik, MD, Principal Investigator — Department of Psychiatry, RSCM
Locations (1):
- Department of Psychiatry, Faculty of Medicine, Universitas Indonesia, Cipto Mangunkusumo National Hospital Jakarta, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
research protocols, analysis

REFERENCES:
- [Background] Kubera KM, Barth A, Hirjak D, Thomann PA, Wolf RC. Noninvasive brain stimulation for the treatment of auditory verbal hallucinations in schizophrenia: methods, effects and challenges. Front Syst Neurosci. 2015 Oct 12;9:131. doi: 10.3389/fnsys.2015.00131. eCollection 2015. PMID 26528145
- [Background] Ray P, Sinha VK, Tikka SK. Adjuvant low-frequency rTMS in treating auditory hallucinations in recent-onset schizophrenia: a randomized controlled study investigating the effect of high-frequency priming stimulation. Ann Gen Psychiatry. 2015 Feb 15;14:8. doi: 10.1186/s12991-015-0046-2. eCollection 2015. PMID 25699086
- [Background] Moseley P, Fernyhough C, Ellison A. Auditory verbal hallucinations as atypical inner speech monitoring, and the potential of neurostimulation as a treatment option. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2794-805. doi: 10.1016/j.neubiorev.2013.10.001. Epub 2013 Oct 12. PMID 24125858